CLINICAL TRIAL: NCT06579456
Title: FormaldEhyde-free embalmeD Cadavers as a Training Tool in a mUltimodal Structured Curriculum in Laparoscopic SURGERY: a Randomized Clinical Trial
Brief Title: Evaluation in a Multimodal Structured Curriculum of Laparoscopic Surgery
Acronym: EDU-SURGERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Los Andes, Columbia (Other)
Responsible Party: Principal Investigator, Roberto Rueda, Associate Professor, University of Los Andes, Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019102254
Record Dates: First submitted 2024-08-20; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Medical Education; Laparoscopic Surgery
Keywords: Laparoscopic Surgical Training; General Surgery; General Surgery Residents; Technical Skills

STUDY DESIGN:
Intervention Model Description: A single-center, single-blind, randomized educational intervention clinical trial was carried out to compare the use of formaldehyde free solution cadaver training in laparoscopic surgery with other traditional simulation surgery options. The trial was approved by our Institutional Research Board, prior to the beginning of the study (Act. No.201910224). Written informed consent was obtained from each participant and the CONSORT statement was followed.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- - Negative control (Active Comparator): participants who continued after the pre-test in this model (negative control group) proceeded with training in the described skills, adding suture training using a perforable MMA-type woven fabric
  Interventions: Other: Negative Control
- - Positive control (Active Comparator): simulation in silicone models was conducted using models that emulate the rigidity, structure, dimensions, and haptic feedback of the anatomical structures to be treated, specifically a hollow viscus for enterorrhaphy training. Each model was placed inside a Pelvitrainer for training, and the participants performed cutting and suturing exercises freely for the allotted time
  Interventions: Other: Positive Control
- Intervention Group (Experimental): training in the cadaveric model was carried out using a complete human body preserved in formaldehyde-free solution. The cadaver was positioned and covered with surgical drapes in the supine position and a pneumoperitoneum was performed for training using a Mindray HD3 laparoscopy tower
  Interventions: Other: Surgical Training Intervention

INTERVENTIONS:
Other: Surgical Training Intervention — Validation of a Formaldehyde-Free embalmed cadavers for recreate with more precision the experience of learning surgical endoscopy
  Arms: Intervention Group
Other: Positive Control — training in models that emulate the rigidity, structure, dimensions, and haptic feedback of the anatomical structures to be treated.
  Arms: - Positive control
Other: Negative Control — Training proceeded in the rigid described skills acquisition platform, adding suture training using a perforable MMA-type woven fabric
  Arms: - Negative control

SUMMARY:
Development of Laparoscopic surgery skills for general surgery residents are considered competencies of major importance. Different tools are used for this purpose, including synthetic models, virtual reality, animal models and human cadaveric specimens preserved by freezing.Cadaveric models share the anatomical similarity, however have some clear disadvantages including the biological risk and the alteration of the mechanical properties of the bodies preserved by this technique, such as tissue rigidness, lack of elasticity and consistency, and the impossibility of achieving adequate pneumoperitoneum. However, we previosly devoleped a formaldehyde free solution for anatomical preservation. Hence. we propose a a single-center, single-blind, randomized educational intervention clinical trial. Research participants who meet the inclusion criteria have a theoretical and practical module on the acquisition of skills in laparoscopy and take a pre-test focused on intracorporeal enterorrhaphy. Subsequently, they are randomized by blocks into three groups: Negative Control, Positive Control, and Intervention, continuing their training in skill acquisition models, silicone models, or Formaldehyde-free solution preserved corpses, respectively. Finally they are evaluated with a post-test. Two blind experts will evaluate participants using the GOALS and OSATS scales for laparoscopic surgery.

DETAILED DESCRIPTION:
General surgery residents (GSR) face several challenges throughout their training, including learning and developing laparoscopic surgery skills (LSS). For GSR, who are constantly subjected to training in minimally invasive interventions, which require training in different skills than traditional surgery - such as minimal invasive manual dexterity, two-dimensional spatial perception and positioning different operating tools amongst others - simulation training (ST) plays an important role in the transition of knowledge acquisition and development of technical expertise during surgical training; The main challenge of ST in minimally invasive surgery is to recreate an environment that achieves both the basic physical parameters and provides decision-making experience during surgery, being its final objective mastering the use and location of the instruments to minimize possible errors during real life surgery. Since the inception of the concept of ST several simulation tools have been created to answer the challenges of training, however evidence suggest that frozen human or animal cadaveric models are the most preferred option by GSR.

Cadaveric models, frozen or fresh, share an anatomical similarity with real practice scenario and accurately reflect the characteristics of human tissues and thus are currently ideal for ST and development of (LSS), however, they present clear disadvantages and limitations that make their use difficult, specially the biological risk and the alteration of the mechanical properties of the bodies preserved by this technique, such as tissue rigidness, lack of elasticity and consistency, and the impossibility of achieving adequate pneumoperitoneum. In response to this issue, there are a variety of preservation techniques that do not use formaldehyde or use minimal amounts of this reagent, however these techniques present their own problems, such as elevated costs, complexity, and poor quality of preservation.

In previous work in our lab, a formaldehyde-free solution was developed and presented as a new preservation solution that claims to maintain -to a certain extent- the color, texture, rigidity, and elasticity of the tissues, allowing the clear identification of anatomical structures, and the creation of adequate pneumoperitoneum at representative low pressures for laparoscopic ST (+/- 5mmHg) after multiple tests. The corpses preserved with this solution can be used for surgical simulation, as they preserved the pose no biosafety risks comparable to those of fresh human tissues, can be reused, and pulse arterial flow can be generated by using an external peristaltic pump articulated with the system.

To our knowledge there is no evidence of the use of human cadaveric specimens preserved with formaldehyde free solutions in LSS development, whereby the aim of this manuscript is to evaluate the use of cadaveric specimens preserved with a formaldehyde free preservation solution as an alternative training tool to develop basic LSS and determine the existence of equivalence between this model and two widely used dry training models.

MATERIALS AND METHODS Design A single-center, single-blind, randomized educational intervention clinical trial was carried out to compare the use of formaldehyde free solution cadaver training in laparoscopic surgery with other traditional simulation surgery options. The trial was approved by our Institutional Research Board, prior to the beginning of the study (Act. No.201910224). Written informed consent was obtained from each participant and the CONSORT statement was followed.

Study Population Medical students who completed their general surgery rotation and general surgery residents of any training level were eligible. Recruitment and selection of the participants was carried out by a formal open invitation through email to the General Surgery coordinators of local University Hospitals and Faculties of Medicine; Likewise, a formal invitation was made to the National Association of Scientific Societies of Medical Students Informed consent was given to all interested parties, and the objective and methodology of the study were explained, as well as the implications of their participation. The interested parties who agreed to voluntarily participate signed the informed consent.

Study Groups All participants received a shared training module divided in a virtual theorical phase of 20 minutes and a hands-on training phase in a Dry Simulator using Jacobeaus simulators of the Cut & Stitch ® brand. Three skills were practiced (cutting, suturing, and transferring) and each skill was trained for 20 minutes per participant, alternately with active breaks every 60 minutes until the proposed training time was completed. The shared module finished with a pretest consisting in integrated task simulation of an enterorrhaphy using laparoscopic approach, using pelvitrainer® with a fresh porcine bowel specimen. After all participants completed the shared module, they were randomized divided into Group A (negative control), Group B (positive control) and Group C (intervention). All three groups were exposed to a training program based on three specifics tasks to make it comparable. These tasks were variations of cutting exercises, suturing exercises and transfer exercises, all of them performed using laparoscopic technique. However, different simulators were used in each group.

* Negative control: participants who continued after the pre-test in this model (negative control group) proceeded with training in the described skills, adding suture training using a perforable MMA-type woven fabric, as shown in.
* Positive control: simulation in silicone models was conducted using models that emulate the rigidity, structure, dimensions, and haptic feedback of the anatomical structures to be treated, specifically a hollow viscus for enterorrhaphy training. Each model was placed inside a Pelvitrainer for training, and the participants performed cutting and suturing exercises freely for the allotted time.
* Intervention: training in the cadaveric model was carried out using a complete human body preserved in formaldehyde-free solution. The cadaver was positioned and covered with surgical drapes in the supine position and a pneumoperitoneum was performed for training using a Mindray HD3 laparoscopy tower.

Analysis Subgroups: analysis subgroups were created to enhance control and intervention comparison. These subgroups were defined as follows:

* Totally naive: Defined as participants who, having completed their surgical rotations and acquired a basic level of knowledge in surgery, have had no practical approach or opportunity to train in any minimally invasive procedures.
* Naive group: Medical Students and Undergraduate Interns who, having completed their surgical rotations and acquired a basic level of knowledge in surgery, have had the opportunity to undergo some training in the acquisition of skills in minimally invasive surgery prior to their participation in the study or have participated as assistants in such procedures.
* Intermediate group: General Surgery Residents who, having had the opportunity to undergo previous training and/or surgical assisting, regardless of the time reported in these, do not exceed 50 hours as the primary surgeon in minimally invasive procedures.
* Expert group: Comprised of General Surgery Residents who, as trainee physicians and regardless of reported training time or assisting, have exceeded 100 hours of acting as the primary surgeon in minimally invasive procedures.

Subgroups were randomly assigned to all three arms including negative control, positive control and intervention.

Design of the Pre-test and Post-test Each test was composed of a predetermined evaluation space in which the participant must perform the simulation of an intracorporeal enterorrhaphy with the support of another participant as an assistant, which was recorded and evaluated according to the Objective Structured Assessment of Technical Skills (OSATS), and the Global Operative Assessment of Laparoscopic Skills (GOALS). Pre-test was defined as the evaluation phase in which participant had only accessed the first shared module. Post-test was defined as the evaluation after randomization. Prior to each test, fresh porcine viscera were assembled inside a pelvitrainer like those used during the training phases, the predisposed trocars were provided, and the instruments were provided next to the pelvitrainer without labels or additional identification marks on the piece. The Mindray HD3 tower laparoscopy camera with 30-degree lens was used.

Masking and Randomization Techniques A single-blind randomized trial was carried out. Participants were included consecutively in groups with a maximum of 6 people for each intervention date. When each participant was included, an anonymous code was assigned to each person, which was then used for identification in the tests, allowing the linking of the results of each pre-test and post-test video. This allows the subsequent analysis of blinded and categorized data according to the level of training and/or anonymous sociodemographic variables obtained from the surveys carried out at the beginning of the study.

Randomization was performed in blocks of 6 in a 2:2:2 ratio using a sealed envelope that contained the intervention or control in which they would participate after taking the pre-test, this process was carried out by an external researcher. The envelopes were prepared by a third party in blocks of 6 each two of them containing one of the three interventions and were previously randomized before being handed out. Inside the envelopes was a piece of paper with the assigned intervention, carbon paper and aluminum paper to prevent anyone from reading the contents when backlit. Before opening the envelope both the participants and one of the researchers signed it, and due to the carbon paper, the sheet with the intervention was signed as well. The participant had no previous knowledge of the information consigned in the envelope and after that, he/she carried out the assigned activities and a post-test.

After capturing the data all test videos were blinded by participant, date, and type (pre-test or post-test) by assigning a 4-digit code generated randomly using the randomize tool between a number less than 1,000 with the command =random.between (=randombetween) from Excel, created and assigned specifically for this study by a third party investigator that would capture and analyze the data. These codes were the only information available to the two evaluators who tabulated the GOALS and OSATS scores ensuring blinding in the analysis. After the assignment of the code and masking the videos, the evaluators were given a password-restricted access folder in a subfolder of OneDrive "Personal Vault", hosted in an institutional Outlook account to access the videos identified with said code.

Outcomes

* Primary Outcome: the main outcome variable assessed was the improvement in Skills in Laparoscopic Surgery evaluated by the difference between the summative score on the GOALS and OSATS scales obtained by the participant between the pre-test and post-test for intracorporeal enterorrhaphy.
* Secondary Outcomes: sociodemographic or dependent variables of the subject were collected, including age, sex, academic post-grad year or medical school year. Variables dependent on the subject's previous training included previous official training in laparoscopy, defined as having taken a course and/or diploma in certified laparoscopy skills training; having carried out surgical assistantships in laparoscopy, defined as support work during laparoscopic surgical procedures as a second surgeon or having helped with the laparoscopic camera during the procedure; and whether they had performed laparoscopic surgical procedures as first surgeon.

Statistical analysis The minimum detectable difference in the assessment and validation scales used was employed to obtain a sample size of n=37 study participants. Inter-observer variability was assessed by means of a concordance test with Cohen's kappa coefficient, however, due to the characteristics of the data collected, a Bland-Altmann difference test (difference plot) was required. Evaluation of the comparability of the two variables was done using the final score of each pre-test and comparing it with other pre-test, as well as comparisons between the pre-test and post-test for each participant and the weighted value for the pre-test vs the weighted value for the post-test.

Subsequently, a comparative analysis was carried out between the three groups (negative control, positive control and intervention) to assess whether they are comparable. Finally, a principal element analysis (PEA) was carried out, discriminating the analysis by educational level, previous training level and possible confounding variables. All analysis were performed using the STATA 17, R and Pas tools, available on the servers of our University.

ELIGIBILITY:
Inclusion Criteria:

1. Fourth, fifth or sixth year medical students over 18 years old who completed their general surgery rotations
2. General Surgery residents over 18 years old at any level of training Over 18 years old.

Exclusion Criteria:

1. Serious illnesses that affect the hability of the participant to safety and ability to complete the study.
2. Participants who have known allergies to components of the interventions or have experienced severe adverse reactions in the past will be excluded from the study.
3. Participants who cannot provide valid informed consent due to cognitive issues, mental impairment, or legal incapacity will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Improvement in Skills in Laparoscopic Surgery using global operative assessment of laparoscopic skills (GOALS) scale | 48 hours
  Pre- and post-intervention individual measures will be taken using the operative assessment of laparoscopic skills (GOALS) to compare the efficacy of the simulated program. The unit of measure are the points of GOALS Scale with a minum score of 5 and a maximum of 25 points. A higher score means a better outcome.
Improvement in the Objective Structured Assessment of Technical Skills (OSATS) global rating scale | 48
  Pre- and post-intervention individual measures will be taken using the Objective Structured Assessment of Technical Skills (OSATS) Scale to compare the efficacy of the simulated program. The unit of measure are the points of OSATS Scale with a minum score of 4 points and a maximum of 20 points. A higher score means a better outcome.

SECONDARY OUTCOMES:
The efficacy given by the progression through the different multimodal methods at OSATS Scale | 48 hours
  The results of the 3 arms will be compared. The unit of measure are the points of OSATS Scale, with a minimum of 4 points and a maximum of 20 points. A higher score means a better outcome.
The efficacy given by the progression through the different multimodal methods at GOALS Scale | 48 hours
  The results of the 3 arms will be compared. The unit of measure are the points of GOALS Scale, with a minimum of 5 points and a maximum of 25 points. A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de los Andes School of Medicine, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No